CLINICAL TRIAL: NCT07387263
Title: Mainstreaming Genetics: Evaluation of a Digital Application to Scale and Spread Oncologist-initiated Genetic Testing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 4066
Record Dates: First submitted 2025-12-17; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Breast Cancer; Prostate Cancer; Colon Cancer; GI Cancers; Ovarian Cancer; Pancreatic Cancer
Keywords: Cancer Genetic Testing; Randomized Controlled Trial; Digital Tool; Mainstreaming; Genetic counseling; Cancer; Genetic testing; Service Delivery; Alternative service delivery model
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm - GA-Mainstream tool users (Experimental): Participants in the intervention arm will use the GA-Mainstream digital tool for cancer genetics education, providing cancer medical and family history, and to support the delivery of their genetic test results. This tool will be used to supplement usual care. Participants will continue to be supported by existing consultations with genetics professionals to discuss their results.
  Interventions: Behavioral: Genetics Adviser for Mainstream Care (GA-Mainstream); Behavioral: Mainstreaming Standard of Care
- Mainstreaming Standard of Care (Active Comparator): Participants in the control arm will receive mainstream care as outlined by the clinic where the patient is being seen, which consists of a patient pamphlet, video and/or a clinician checklist for pre-test counseling. Results will be disclosed by either a genetic counselor or oncologist with post-test counseling of select patients.
  Interventions: Behavioral: Mainstreaming Standard of Care

INTERVENTIONS:
Behavioral: Genetics Adviser for Mainstream Care (GA-Mainstream) — The Genetics Adviser for Mainstream Care will educate participants on cancer genetic testing after oncologist-initiated genetic testing. Participants may also receive their results on the GA-Mainstream.
  Other Names: GA-Mainstream
  Arms: Intervention arm - GA-Mainstream tool users
Behavioral: Mainstreaming Standard of Care — After oncologist-initiated genetic testing, participants may not receive additional information prior to the receipt of their results or they may receive educational materials on cancer genetic testing. Results will be disclosed by either a genetic counselor or oncologist with post-test counseling of select patients.

SUMMARY:
Genetic testing can alter therapy and surgical management for cancer patients and is therefore indicated as a first-line test for many newly diagnosed patients, including breast, ovarian, pancreatic, prostate and colon/GI patients. To reduce pressure on already constrained genetics clinics across Canada, some cancer centres are 'mainstreaming' genetic testing - whereby genetic testing is initiated and mediated by oncologists without traditional pre-test genetic counseling (GC) often using some form of paper-based patient pamphlets or videos. There is no standard, evidence-based approach to mainstreaming, leading to significant practice variation, a lack of coordinated care and ultimately, negative psychological impacts on patients. Digital solutions can address these gaps by providing a standardized, coordinated and patient-centered approach to deliver cancer genetic education. However, digital solutions for providing cancer genetics services are uncommon and clinical-effectiveness and service delivery outcomes have not been well-assessed. This study will test a digital mainstreaming platform called the Genetics Adviser for Mainstream care to assess its effectiveness in improving psychological outcomes and patient-centred care for mainstream cancer patients compared to standard of care.

DETAILED DESCRIPTION:
Background: Germline genetic testing can alter therapy and surgical management for cancer patients. Yet, the rising demands for genetic testing and counseling has added pressure to already constrained genetic counseling (GC) service models that require extensive pre-test GC with a genetic counselor. Many cancer genetics centres are 'mainstreaming' genetic testing, replacing traditional pre-test GC, where genetic testing is initiated and mediated by oncologists, using clinician checklists, patient pamphlets, or videos. Most evidence on cancer genetics mainstream models to date derives from uncontrolled, non-randomized studies with limited outcomes. Electronic patient portals and digital decision tools have been shown to improve psychological outcomes.

Rationale: There is no standard, evidence-based approach to 'mainstreaming', leading to significant practice variation, a lack of coordinated care and ultimately, negative psychological impacts on patients. Digital solutions can address these gaps by providing a standardized, coordinated and patient-centred approach to deliver cancer genetic counseling. This study will address these gaps by testing the effectiveness of the Genetics Adviser for Mainstream Care (GA-Mainstream), building on our rigorously-evaluated digital health application called the Genetics Adviser.

Primary Objective: Assess the clinical effectiveness of the GA-Mainstream in improving psychological outcomes (e.g. test-specific distress), and patient-centred care (e.g. knowledge, and empowerment) for mainstream cancer patients compared to those receiving standard mainstream care.

Secondary Objectives:

* Measure the impact of the GA-Mainstream on patients' risk perceptions and intent to follow clinical recommendations (e.g. surveillance, treatment changes, or cascade testing).
* Assess efficiencies in turnaround time to test result disclosure and time spent in genetic counselling sessions between groups.
* Understand the experiences of patients and providers with the GA-Mainstream and the process of receiving genetic testing results through the platform.

Hypotheses

* Patients who use the GA-Mainstream will report lower distress and higher knowledge and empowerment compared to standard-of-care mainstream patients.
* Patients using the GA-Mainstream will have more accurate risk perceptions and higher intent to follow clinical recommendations.
* Using the GA-Mainstream will reduce turnaround time and increase efficiency during genetic counselling sessions.

Methods: This is a mixed-method, non-blinded randomized controlled superiority trial. The trial will evaluate whether the use of the GA-Mainstream reduces test-specific distress compared to standard mainstream genetic testing. As part of this trial, patients will receive germline genetic testing.

Study Population: Adult patients (aged >18 years) referred for mainstream cancer genetic testing related to ovarian, pancreatic, breast, prostate, or GI cancers.

Sample Size: Our primary outcome, test-specific distress measured using the MICRA, has an accepted minimal clinically important difference (MCID) of 2.5. Assuming this, 64 participants/arm (128 total) are estimated to be required to have 80% power at a 2-sided significance level of 0.05 to detect the MCID using a standard two-sample t-test.

Intervention: Participants in the intervention arm will use the GA-Mainstream to support the delivery of their genetic test results, including collecting cancer medical history and family cancer history, pre- and post-result education. The GA-Mainstream will supplement mainstream standard of care.

Control: Participants in the control arm will receive standard of care for mainstream patients as outlined by the clinic where the patient is being seen, which consists of a patient pamphlet, video, or clinician checklist for pre-test counseling and results disclosure by either a genetic counselor or oncologist with post-test counseling of select patients.

Primary Outcome: The primary outcome is test- specific distress, measured by the Multidimensional Impact of Cancer Risk Assessment (MICRA).

Secondary Outcomes: Generalized distress, measured by the Hospital Anxiety and Depression Scale (HADS); Knowledge, measured by the KnowGene questionnaire; empowerment, measured by the Genomics Outcome Scale (GOS-6); Self-efficacy, measured by the Genetic self-efficacy scale; Quality of life measured by the 12-item Short Form Health Survey (SF-12); Satisfaction with genetics education and intended health behaviour change, assessed by team developed questions; Satisfaction with digital tool measured by the Digital Health Application Satisfaction Scale (DHASSP); digital health literacy measured by digital health care literacy scale; health literacy measured by the BRIEF Health Literacy Screening tool.

Turnaround times will be measured by documenting time between blood draw, return of result and result disclosure by the clinician. Time saved will be measured by capturing time spent preparing for the session, during the session with the genetic counselor, and after the session across both arms. Frequency of platform use will also be documented and duration of platform use by recording platform access dates and time.

Quantitative Analysis: Analysis will follow the intention-to-treat approach. Mean scores for test-specific distress will be compared using a t-test. Secondary outcomes of generalized distress, empowerment, and knowledge will also be analyzed using a t-test for hypothesis-generating purposes; therefore no multiplicity corrections will be applied. Mean wait times, total consult times and frequency and duration of use between arms will be analyzed descriptively and compared using a t-test. P-values will be set at 0.05 (two-tailed).

Qualitative Study: Following the trial, qualitative interviews will explore users' experiences with the GA-Mainstream. This will be used to explore participants' experiences, perceptions, and needs related to the use of the GA - Mainstream platform. A purposeful sample of study participants will be used. A mix of intervention arm participants (n=30) will be identified across cancer type, result type, and demographic characteristics to assess patient experience using the GA-Mainstream.

Qualitative Analysis: The qualitative analyses will draw on an interpretive description approach, using open coding and constant comparison to identify common and divergent themes. Interviews will consider participants' socio-demographic factors that may influence their informational and decisional needs, as well as how they engage with genetic information and participate in shared decision making. Two researchers will code transcripts independently; consensus on codes will be reached through discussion. Ongoing analysis will inform the development of progressive iterations of the interview guides.

Mixed-Methods Integration: The quantitative and qualitative data will be integrated to understand whether the tool is effective, including how and why it may influence outcomes such as distress, empowerment, and risk perception. Quantitative and qualitative findings will be narratively described and integrated using a convergent design matrix and joint displays, merged if appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Receiving germline testing related to primary cancer condition initiated by oncologist
* 18 years old or older.
* Speak and read English

Exclusion Criteria:

* Receiving cancer genetic testing via a referral to a genetics clinic
* Do not speak or read English
* Under 18 years of age
* Determined to have diminished, marginal and or fluctuating decisional capacity
* Lack access to internet or an electronic device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Test Specific Distress - Multi-Dimensional Impact of Cancer Risk Assessment (MICRA) | Assessed immediately after return of results via intervention (intervention arm only). Assessed at 2-weeks (primary timepoint) and 6 weeks post-return of results for everyone.
  The Multi-Dimensional Impact of Cancer Risk Assessment (MICRA) is a 25-item standardized, validated scale that measures the impact of result disclosure from genetic tests. There are three subscales: Distress (6 items), Uncertainty (9 items) and Positive Experiences (4 items). Total scores range from 0-125, with higher scores indicating worse outcome. Scores on the Distress subscale range from 0-30, with higher scores indicating worse outcome. Scores on the Uncertainty subscale range from 0-45, with higher scores indicating worse outcome. Scores on the Positive Experiences Subscale range from 0-20, with higher scores indicating worse outcomes. (PMID: 12433008)

SECONDARY OUTCOMES:
Generalized Distress - Hospital Anxiety & Depression Scale (HADS) | Assessed at all timepoints: a)Baseline; b) 3-weeks after baseline; c) 2-weeks post-return of genetic test results; and d) 6-weeks post-return of results. Intervention arm only: e) Post first digital tool use, & f) post-return of results via intervention.
  The Hospital Anxiety and Depression Scale (HADS) is a validated tool that assesses symptoms of anxiety and depression in medical and general populations. It consists of 14 items divided into two subscales: Anxiety (HADS-A) and Depression (HADS-D), each with 7 items scored on a 4-point Likert scale with scores ranging from 0-21 per subscale. The measure captures generalized psychological distress by evaluating non-somatic symptoms, making it suitable for use in clinical settings where physical illness may confound mood assessment. Higher scores indicate greater severity of anxiety and depressive symptoms, with established cut-offs for mild, moderate, and severe distress.
Knowledge - KnowGene | Assessed at all timepoints: a)Baseline; b) 3-weeks after baseline; c) 2-weeks post-return of genetic test results; and d) 6-weeks post-return of results. Intervention arm only: e) Post first digital tool use, & f) post-return of results via intervention.
  Knowledge will be measured using KnowGene, a measure of knowledge about cancer genetic after cancer genetic counseling and multigene panel testing, an effective and established 16-item questionnaire. Response options include: agree, disagree, or 'don't know'. Either agree or disagree was considered a correct response, depending on the item, with responses being assigned a value of 0 or 1. Higher knowledge scores indicate a higher level of knowledge.
Empowerment - Genomics Outcome Scale (GOS-6) | Assessed at all timepoints: a)Baseline; b) 3-weeks after baseline; c) 2-weeks post-return of genetic test results; and d) 6-weeks post-return of results. Intervention arm only: e) Post first digital tool use, & f) post-return of results via intervention.
  Measured by the Genomics Outcome Scale (GOS-6). The Genomics Outcome Scale (GOS) is a 6-item scale that measures empowerment and is a validated short-form of the 24-item Genetic Counselling Outcome Scale (GCOS-24). The 6-item GOS is shorter and more broadly applicable, such as in circumstances where a non-genetics provider has disclosed a result or when results are disclosed online. The GOS includes a 5-point Likert scale from strongly disagree (1 point) to strongly agree (5 points) for a possible score range of 6-30 points on this scale. (PMID: 30496830)
Self-Efficacy - Genetic Self Efficacy Scale | Assessed at all timepoints: a)Baseline; b) 3-weeks after baseline; c) 2-weeks post-return of genetic test results; and d) 6-weeks post-return of results. Intervention arm only: e) Post first digital tool use, & f) post-return of results via intervention.
  Measured by the Genetic Self Efficacy scale. This 5-item scale measures individuals' confidence in their ability to understand the genetic information provided. Participants will be asked to indicate their level of agreement or disagreement (7-point Likert scale from 1 = strongly disagree to 7 = strongly agree). Responses to the items will be summed, with higher scores indicating greater self-efficacy (range: 5-35).
Quality of Life - Short Form Health Survey (SF-12) | Assessed at baseline, 2 weeks post return of results (primary timepoint), and 6 weeks post return of results.
  Quality of life will be measured using the Short Form Health Survey (SF-12). This 12-item scale captures physical and mental health providing a physical component summary and mental component summary to capture health on the individual level. The SF-12 uses a 4-week recall period and is sensitive to changes in health over time.
Satisfaction with Genetics Education | Assessed at all timepoints: a)Baseline; b) 3-weeks after baseline; c) 2-weeks post-return of genetic test results; and d) 6-weeks post-return of results. Intervention arm only: e) Post first digital tool use, & f) post-return of results via intervention.
  Satisfaction with genetics education will be assessed using items adapted from PMID: 28791521. Participants will rate clarity, helpfulness, and overall satisfaction with the education format using Likert-scale questions (e.g., 1 = very dissatisfied to 5 = very satisfied). Scores will be summed, with higher scores indicating greater satisfaction.
Risk Perception - TRIpartite model of RISK perception (TRIRISK) | Assessed at a) Baseline; b) 2-weeks post-return of genetic test results; and c) 6-weeks post-return of results. As well as immediately after the return of results via intervention (intervention arm only).
  Risk perception will be measured by the Tripartite Model of Risk Perception (TRIRISK), an 18 item scale assessing deliberative, affective, and experiential perceptions. These components are used to understand how people perceive and react to different health and other risks. Items are scored using 7-point Likert scales or percentage ratings. Each subscale has six items, and scores are averaged within each domain for a total score of 126. A high deliberative score means the person logically believes they are at high risk (e.g., based on probability). A high affective score means they feel emotionally concerned or worried about the risk. A high experiential score means they intuitively or personally feel vulnerable to the risk.
Intended Health Behavioural Change Questions | Assessed at a) baseline, b) 3-weeks after baseline; c) immediately after viewing results via the platform (intervention only), d) 2-weeks post-return of results, and e) 6-weeks post-return of results.
  Guided by the health belief model of behaviour change, six questions were developed by the research team guided by the literature and experts. Questions will inquire about participants' intentions to: 1) obtain more information, 2) share genetic results with family, 3) communicate results with healthcare providers, 4) make lifestyle changes, 5) pursue screening, and 6) have preventative surgery.
Satisfaction with Digital Tool - Digital Health Application Satisfaction Scale (DHASSP) | Administered to the intervention arm only immediately post-intervention, after the return of results via intervention, and at 2 weeks post-return of results.
  Measured using the Digital Health Application Satisfaction Scale (DHASSP) to capture satisfaction with the digital tool, including usability, perceived usefulness, ease of navigation, and overall experience. Items are rated on a Likert scale (strongly disagree to strongly agree), with higher scores indicating greater satisfaction. The scale provides insight into user engagement and acceptability of the digital intervention.

OTHER OUTCOMES:
Qualitative interviews with a subset of participants and providers | 1-6 months following return of results.
  Interviews with patients will be used to gain further insights into the delivery and support of mainstreaming genetic services with the support of a digital intervention.
Health Literacy - BRIEF | Assessed at baseline.
  Health literacy will be assessed using the BRIEF Health Literacy Screening Tool, a 4-item measure designed to identify an individual's ability to understand and use health information. Each item is quantified using a 5-point scale (1-5) with higher scores indicating higher health literacy.
Digital Health Literacy - Digital Health Care Literacy Scale | Assessed at baseline.
  Measured by the Digital Health Care Literacy Scale, a 3-Item measure of digital health literacy. Each item uses a 5-point Likert scale to answer each question with response options ranging from "strongly agree" (4 points) to "strongly disagree" (0 points). The sum of individual items is used to create the total score. Possible scores range from 0 to 12, with higher scores indicating higher digital health care literacy skills.
Clinician time preparing for the session, counseling and post-session | Collected at 2-weeks post-test result disclosure by the clinician.
  Measure of total time spent preparing for the genetic counselling session, time with the Genetic Counselor in the counselling session and time spent preparing letters and chart notes after the session. Collected for both the intervention and control arm.
Efficiency - Turnaround time | Collected at 2-weeks post-test result disclosure by the clinician.
  To capture any efficiency caused by the intervention, turnaround time will be measured by collecting the date of blood draw, the date the genetic test report was returned, and the date of disclosure (by intervention vs. by clinician).
Frequency of platform use | Collected at the end of participation in the study at 6-weeks post-test result disclosure (intervention arm only).
  Measure of the number of times the digital platform was accessed by the participant. Intervention arm only.
Duration of platform session | Collected at the end of participation in the study at 6-weeks post-test result disclosure (intervention arm only).
  Measure of total time spent per participant using the digital platform. Intervention arm only.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Bombard, PhD, Principal Investigator — St. Michael's Hospital and University of Toronto
Locations (2):
- Canada (2):
  - Sunnybrook Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to research who are interested in / conducting similar research in this field. This data will be available upon request, keeping with research ethics procedures.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Data will be made available to research who are interested in / conducting similar research in this field. This data will be available upon request, keeping with research ethics procedures.
URL: https://oldresearch.unityhealth.to/labs/yvonne-bombard/